CLINICAL TRIAL: NCT02409797
Title: measurINg forceS durInG cHiropractic Treatment (INSIGHT): A Single-Arm Clinical Case Series
Brief Title: measurINg forceS durInG cHiropractic Treatment
Acronym: INSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INSIGHT-2015V164
Record Dates: First submitted 2015-03-12; First posted 2015-04-07 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flexion-Distraction spinal manipulation (Experimental): Participants will receive Flexion-Distraction treatment from a licensed doctor of chiropractic. During the procedure the participant lies prone on a specially designed treatment table. The table is equipped with a movable lower body section, which can be directed by the study doctor to lower the participants legs, move them from side to side, or in a traction motion. Table movements can occur in combination with other motions, depending on the diagnosis and characteristics specific to the participant's condition. During this procedure, the doctor will also touch the lower or upper part of the participants back or neck with their hands to direct treatment toward specific spinal regions.
  Interventions: Other: Flexion-Distraction (non-thrust) spinal manipulation

INTERVENTIONS:
Other: Flexion-Distraction (non-thrust) spinal manipulation — Enrolled participants will receive chiropractic care over a 2-week period. Chiropractic care includes standard therapies for back pain. A doctor of chiropractic determines the therapeutic approach and treatment frequency based upon a participant's clinical presentation. If provided, treatments will include low-velocity (non-thrust) spinal manipulation using the Flexion-Distraction procedure. Recommendations for exercise, lifestyle modifications, or other therapies may also be provided.

SUMMARY:
The INSIGHT pilot study will measure forces applied by a doctor of chiropractic (DC) during the delivery of a specific, manually based chiropractic treatment for participants with low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is a well-recognized health problem. One common manual therapy available for the treatment of LBP is spinal manipulation (SM), which can be separated into 2 categories: High-Velocity Low-Amplitude (thrust) and Low-Velocity (non-thrust) SM according to their force-delivery profiles. One commonly utilized non-thrust SM technique is the Flexion-Distraction procedure. Several studies have reported manually applied forces during thrust SM; however, the forces used during non-thrust SM, specifically those used with Flexion-Distraction treatment are still unknown. The results of this pilot study will provide preliminary information on treatment forces and sample size justification for future full-scale trials, while also ascertaining the feasibility of the study protocol and patient recruitment methods for such trials.

ELIGIBILITY:
Inclusion Criteria:

* Able to demonstrate the necessary abilities (English language, literacy) needed to provide informed consent without the assistance of another person (e.g., a proxy, spouse, family member or other support person)
* Self-reported low back pain (acute, subacute or chronic) at the time of examination and enrollment

Exclusion Criteria:

* Weight > 300lbs
* Spinal Pathology or conditions contraindicating study procedures or compromising participant safety
* Inflammatory arthropathy involving the spine (e.g. Ankylosing spondylitis, Rheumatoid arthritis)
* Spinal fracture in the past 6 months
* Other conditions requiring referral (e.g. self-reporting alcohol/substance dependence or abuse, unstable spinal segments, and cauda equina syndrome)
* Pregnant or planning to become pregnant within the next 5 weeks
* Unable to tolerate study procedures safely
* Altered Mental Capacity
* Sensitivity to adhesives used in the study
* Uncontrolled hypertension
* Co-morbidity requiring simultaneous clinical management that compromises ability to deliver study procedures or assess the participant's heath status or poses as a scheduling burden
* Retention of legal advice or seeking a health-related insurance claim
* Compliance concerns (e.g. scheduling conflicts, moving from the quad city area, unwilling to undergo required study procedures or receive treatment from study doctor(s))
* Quebec Task Force Classification of 10 or 11: (chronic pain syndrome, visceral/infectious source of LBP)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Traction forces | Baseline and 2 weeks
  We will measure traction forces delivered to the participant by the clinician during all study visits over a 2-week time period. Traction forces will be summarized descriptively with means and standard deviations. Primary outcomes will compare changes in traction forces between the baseline and final treatment visit at 2 weeks.

SECONDARY OUTCOMES:
Pain Visual Analog Scale (VAS) | Baseline and 2 weeks
  The Visual Analog Scale (VAS) will be used to assess the participant's current back pain level and their average back pain levels over the past 24hrs and week. Participants will be asked to rate their level of pain on a 100 millimeter continuum horizontal scale with no pain and worst imaginable pain anchors.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Vining, DC, Principal Investigator — Palmer Center for Chiropractic Research (PCCR)
Locations (1):
- Palmer Center for Chiropractic Research, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Feasibility/pilot study